CLINICAL TRIAL: NCT00644878
Title: A Multi-center, Open-label, Exploratory Study of Bcr-Abl Kinetics in Adult Patients on Nilotinib With Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP) and a Suboptimal Molecular Response to Imatinib
Brief Title: Study of Molecular Response in Adult Patients on Nilotinib With Philadelphia Chromosome Positive Chronic Myelogenous Leukemia (Ph+ CML) in Chronic Phase and a Suboptimal Molecular Response to Imatinib
Acronym: MACS0254
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slower than expected enrollment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107AUS09
Record Dates: First submitted 2008-03-19; First posted 2008-03-27 (Estimated); Results first posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Chronic Myelogenous Leukemia - Chronic Phase
Keywords: leukemia; chronic myelogenous leukemia; chronic phase; molecular response; nilotinib; ENABL
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nilotinib (Experimental)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib 300 mg is taken by mouth twice a day at 12 hour intervals. Nilotinib is to be taken with water on an empty stomach. No food two hours prior to the dose of nilotinib and for one hour following the dose.
  Other Names: Tasigna; AMN 107

SUMMARY:
This exploratory study will evaluate the change in molecular response in chronic myelogenous leukemia - chronic phase patients with a complete cytogenetic response and have a suboptimal molecular response to imatinib

ELIGIBILITY:
Select Inclusion Criteria:

* Male or female patients ≥ 18 years of age with a confirmed diagnosis of Ph+ CML-CP and CCyR
* A suboptimal molecular response to imatinib defined as:

  * Group 1: Treated with 1 year of imatinib, complete cytogenetic response (CCyR) but no major molecular response (MMR) (Bcr-Abl levels >0.1%IS);
  * Group 2: No specific duration of imatinib required, achieved CCyR but has >1 log increase in Bcr-Abl transcript levels
* Adequate end organ function
* Patients must have had an imatinib washout period of at least 3 days and not to exceed 7 days prior to the first dose of nilotinib. Group 1 patients must have been treated with imatinib for at least 1 year. There was no imatinib treatment duration requirement for Group 2 patients.
* For Group 1, patients were eligible for screening if they were treated with an imatinib dose of at least 400mg daily. Dose reduction could have occurred as long as the minimum dose was 300mg daily and the reduction lasted ≤ 28 days. The patient was required to be on 400 mg daily (or a higher dose) of imatinib for at least 6 consecutive months leading up to screening for this study.
* For Group 2 patients, dose reduction while on imatinib could have occurred as long as the minimum dose was 300 mg daily, and the reduction lasted ≤28 days.

Select Exclusion Criteria:

* Prior accelerated phase or blast crisis CML
* Patients achieving prior CCyR on imatinib who lost cytogenetic response prior to entering study
* Previously documented T315I mutations
* Prior therapy with any other tyrosine kinase inhibitor except imatinib
* Patients with contraindications to receiving nilotinib, including concomitant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (11):
  - USC Norris Cancer Center Jane Anne Nohl, Los Angeles, California
  - Georgia Health Sciences University Dept. of MCG, Augusta, Georgia
  - Indiana Blood and Marrow Institute, Beech Grove, Indiana
  - University of Iowa Hospitals & Clinics Univ of Iowa Hosp & Clinic, Iowa City, Iowa
  - LSU HEALTH SCIENCES CENTER/ LSU SCHOOL OF MEDICINE Feist-Weiller Cancer Center, New Orleans, Louisiana
  - St. Agnes Hospital, Baltimore, Maryland
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - South Texas Institute of Cancer, Corpus Christi, Texas
  - Baylor College of Medicine - Breast Care Dan L Duncan Cancer Ctr, Houston, Texas
  - Central Utah Clinic Central Utah Clinic (7), Provo, Utah
  - Froedert Memorial Lutheran Hospital Dept.ofFroedert Memorial, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Ailawadhi S, Akard LP, Miller CB, Jillella A, DeAngelo DJ, Ericson SG, Lin F, Warsi G, Radich J. Exploratory study on the impact of switching to nilotinib in 18 patients with chronic myeloid leukemia in chronic phase with suboptimal response to imatinib. Ther Adv Hematol. 2017 Jan;8(1):3-12. doi: 10.1177/2040620716678118. Epub 2016 Nov 24. PMID 28042454

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 12 centers in United States.
Pre-assignment Details: A total of 18 participants was enrolled in this study. Due to slower than expected enrollment, the study was terminated on 31 March 2012.
Groups:
- Nilotinib: Participants orally received a total of 600 milligram (mg) dose of Nilotinib as 50-mg and 200-mg hard gelatin capsules twice daily (BID) for 12 cycles (each cycle = 28 days).
Period: Overall Study
Arm/Group | Nilotinib
Started | 18
Completed | 0
Not Completed | 18
Not completed — Adverse Event | 2
Not completed — Abnormal laboratory value | 3
Not completed — Protocol deviation | 2
Not completed — Treatment duration completed as per protocol | 11

BASELINE CHARACTERISTICS:
Population: The analysis was performed in Intent-to-treat (ITT) population, defined as all enrolled participants who received at least 1 dose of study drug and had at least 1 post-baseline assessment.
Groups:
- Nilotinib: Participants orally received a total of 600 mg dose of Nilotinib as 50-mg and 200-mg hard gelatin capsules BID for 12 cycles (each cycle = 28 days).
Arm/Group | Nilotinib
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 14
  Black | 0
  Asian | 1
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Log Change From Baseline in Breakpoint Cluster Region Gene (BCR) - Abelson Proto-oncogene (ABL) (Bcr-Abl) Transcript Levels
Description: The change on a logarithmic scale at 12 months from a standardized baseline value (100% on the international scale [IS]) in Bcr-Abl transcripts as assessed by peripheral blood Quantitative real-time polymerase chain reaction (RQ-PCR).
Time Frame: From Baseline up to 12 Months
Population: The analysis was performed in intent-to-treat (ITT) population, defined as all enrolled participants who received at least 1 dose of study drug and had at least 1 post-baseline assessment. Here, number of participants analyzed refer to the number of participants evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: log change
Arm/Group | Nilotinib
Number analyzed (Participants) | 18
log change
  Baseline | 2.229 (0.6165)
  Month 12: number analyzed (Participants) | 12
  Month 12 | 3.612 (0.5689)

2. Secondary Outcome: Number of Participants Who Achieved Major Molecular Response (MMR)
Description: Major Molecular Response (MMR) value at molecular MD is designated a percentage, which is equivalent to a 3-log reduction from a standardized baseline value from the International Randomized InteYesrferon versus STI571 (IRIS) study or 0.1 percent (%) per International Scale (IS).
Time Frame: From Baseline up to 12 Months
Population: The analysis was performed in ITT population, defined as all enrolled participants who received at least 1 dose of study drug and had at least 1 post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 18
Participants
  Baseline: Response: Yes | 0
  Baseline: Response: No | 18
  Baseline: Response: Missing | 0
  Month 12: Response: Yes | 9
  Month 12: Response: No | 3
  Month 12: Response: Missing | 6

3. Secondary Outcome: Number of Participants Achieved Reduction From a Standardized Baseline Value in Bcr-Abl Transcript Levels up to Month 12
Description: Number of participants experiencing either a greater than or equal to (>or=) 1, >or= 2, or >or= 3 log10 reduction in Bcr-Abl transcript levels from Baseline to End of Cycle (EOC) 45 (Day1219 - Day1302) were presented.
Time Frame: From Baseline up to 12 Months
Population: The analysis was performed in ITT population, defined as all enrolled participants who received at least 1 dose of study drug and had at least 1 post-baseline assessment. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 12
Participants
  >or=1 log10 reduction | 12
  >or= 2 log10 reduction | 12
  >or= 3 log10 | 9

4. Secondary Outcome: Median Time to Best Molecular Response
Description: The median time to best molecular response, defined as the time (in months) from the date of enrollment to the date when the maximum reduction in Bcr-Abl transcript level was observed.
Time Frame: From Start of Study up to End of the Study (up to 41 Months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nilotinib
Number analyzed (Participants) | 18
months | 13.8 [4.2 to 23.1]

5. Secondary Outcome: Duration of Best Molecular Response
Description: Duration of best molecular response, defined as the time (in months) from the date of best molecular response to a date when an increase in >1 log10 was observed
Time Frame: From Start of Study up to End of the Study (up to 41 Months)
Population: Since only one participant met the criterion of losing response (that is [i.e.,] an increase in > 1 log10 is observed after the occurrence of best molecular response), the analysis was not performed. Hence data was not collected and reported.
Arm/Group | Nilotinib
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With an Event-free Survival
Description: Event-free survival was defined as the number of participants from the date of enrollment to the date of first occurrence of any of the following: loss of complete hematological response (CHR), loss of Complete cytogenetic response (CCyR), >1 log increase in Bcr-Abl transcripts from the lowest recorded value, progression to accelerated or blast phase, and death.
Time Frame: From Start of Study up to End of the Study (up to 41 Months)
Population: The analysis was performed in ITT population, defined as all enrolled participants who received at least 1 dose of study drug and had at least 1 post-baseline assessment. Participants who did not have an event or dropped out without an event are considered censored at the date of the last observed event.
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 18
Participants
  Event | 1
  Censor | 17

7. Secondary Outcome: Number of Participants With a Progression-free Survival
Description: Progression-free survival was defined as the number of participants from the date of enrollment to the date of first occurrence of progression to Accelerated phase (AP) or Blast crisis (BC) phase, chronic myelogenous leukemia (CML) or death. Participants who did not have an event or dropped out without an event are considered censored at the date of the last observed event.
Time Frame: From Start of Study up to End of the Study (up to 41 Months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 18
Participants
  Censor | 15
  Missing | 3

8. Secondary Outcome: Number of Participants With an Overall Survival
Description: Overall survival was defined as the number of participants from enrollment to the date of death.
Time Frame: From Start of Study Enrollment up to End of the Study (up to 41 Months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 18
Participants | 18

ADVERSE EVENTS:
Time Frame: From Start of Study to End of the Study (up to 41 Months)
Description: The analysis was performed on safety set population defined as all participants who received study drug and had at least one post-baseline safety assessment.
Groups:
- Nilotinib: Participants orally received a total of 600 mg dose of Nilotinib as a as 50-mg and 200-mg hard gelatin capsules BID for 12 cycles (each cycle = 28 days).
Arm/Group | Nilotinib
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=18)
Bradycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=18)
Anaemia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Dry eye (Eye disorders) | 3
Eye irritation (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Macular degeneration (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Anal pruritus (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Proctalgia (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Fatigue (General disorders) | 6
Irritability (General disorders) | 1
Swelling (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Seasonal allergy (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 4
Tinea infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood magnesium increased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 5
Hyperaesthesia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Loss of libido (Psychiatric disorders) | 1
Bladder prolapse (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Breast tenderness (Reproductive system and breast disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Sexual dysfunction (Reproductive system and breast disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 5
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated on 31 March 2012 due to slower than planned enrollment, resulting in a small sample size, no inferential analyses were conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes